CLINICAL TRIAL: NCT02959346
Title: Investigate the Efficacy of Acupuncture in Postoperative Pain Control for Minimal Invasive Thoracoscopic Surgery Patients
Brief Title: Acupuncture in Postoperative Pain Control for Minimal Invasive Thoracoscopic Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH105-REC2-097
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Acupuncture; Pain Control; Randomized Controlled Trial; Thoracic Surgery
Keywords: Minimal invasive thoracoscopic surgery; Pain control; Acupuncture; Randomized controlled trial
MeSH Terms: conditions — Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Acupuncture (Sham Comparator): After recruitment, participants will be randomized to receive acupuncture or sham acupuncture treatment. In the sham acupuncture group, participants will receive sham acupuncture.
  Interventions: Procedure: Sham Acupuncture
- Acupuncture (Experimental): After recruitment, participants will be randomized to receive acupuncture or sham acupuncture treatment. In the acupuncture group, participants will receive acupuncture.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Sham Acupuncture — Procedure:
  Sham Acupuncture(ipisilateral side, 0.3cun, No needle sensation (de qi) was elicited) Sham acupuncture will be applied by inserting acupuncture needle into acupoints(1cm away from the true acupoint):upper limb: Waiguan TE5; lower limb: Zusanli ST36.
  All procedures were carried out to a depth of 0.5 cm with disposable needles measuring 0.16 mm in diameter (40-gauge) and 12.7 mm in length (Yu Kuang, Taipei, Taiwan).
  Acupuncture treatment will consist of one session per day and consecutive three days after thoracoscopic surgery.
  Arms: Sham Acupuncture
Procedure: Acupuncture — Procedure:
  Acupuncture(ipisilateral side, the needling depth decided by whether patients feel De qi, neutral supplementation and draining) Acupuncture will be applied by inserting acupuncture needle into acupoints: Zhigou TE6, Shousanli LI10, Hegu LI4, Neiguan PC6, Houxi SI3; lower limb: Biguan ST31, Fushe SP13, Zulinqi GB41; axillary area(Remove Needles right away after De qi): Yuanye GB22, Jiquan HT1; local area(Remove Needles right away after De qi): ashi point close to the pain area.
  The other needles will be left for 20 minutes and then removed. All procedures were carried out with disposable needles measuring 0.25 mm in diameter (32-gauge) and 44 mm in length (Yu Kuang, Taipei, Taiwan).
  Acupuncture treatment will consist of one session per day and consecutive three days after thoracoscopic surgery.
  Arms: Acupuncture

SUMMARY:
Minimal invasive thoracoscopic surgery has been used widely for common thoracic diseases in recent years. Patients who received thoracoscopic surgery recovered much quickly and returned to their daily life sooner because of small operation wound and less invasion. However, operative pain was still an important factor, which might contribute to several post-operative complications.

In daily practice, patients received oral/intravenous form non-steroidal anti-inflammatory drugs and opioid agents, or patient-controlled analgesia for post operative pain control. However, some side effects were observed occasionally.

The role of acupuncture in post-operative pain control was frequently discussed in recent research. The main mechanisms of acupuncture in pain control were (1) to stimulate the release of endogenous opioid and (2) to block TRPV1 receptor.

The randomized controlled trial arranged by Gary Deng and his colleagues in 2008, was the first clinical trial investigated the role of acupuncture in post-operative pain control for traditional thoracotomy patients. However, there was no further research about the role of acupuncture applied to minimal invasive thoracoscopic surgery.

Thus, the aim of this randomized controlled trial was to investigate the role of acupuncture in post-operative pain control for minimal invasive thoracoscopic surgery patients. In order to deliver a safe and effective way in pain control, and to save medical cost and promote quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20-year-old
* Both male and female patients
* Nationality: Republic of China (R.O.C., Taiwan)
* Who received thoracoscopic surgery for benign lung tumor/disease, metastatic lung tumor, primary lung cancer, mediastinal tumor

Exclusion Criteria:

* Abnormal function of coagulation
* Platelet count less than 20 x 10^3/mm^3
* International normalized ratio (INR) more than 2.5
* Severe comorbidity, for example central vascular, cardiovascular disease, liver/renal failure
* Who would not cooperate in access, or express appropriately

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain scale at post operative day 2, after intervention | measure at post-operative day 1, 9AM, before intervention; and post-operative day 2, 5PM, after intervention
  1. Pain, as assessed by Numeric Rating Scale, NRS
  2. Measure at post-operative day 1, 9AM, before intervention; and post-operative day 2, 5PM, after intervention
  3. accompanied with rest, deep breath, cough and change posture by left and right decubitus

SECONDARY OUTCOMES:
Opioid dosage | injection times of morphine or ketorolac would be recorded during whole admission, an average of 7 days
  1. Routine pain control was given with oral form acetaminophen (500mg, at every 9AM, 1PM, 5PM and 9PM)
  2. Additional Morphine was given for intolerable pain (0.05mg/kg, intramuscular injection)
  3. Additional Ketorolac was given for intolerable pain after morphine used (15mg, intramuscular injection)
  4. Avoid patient controlled analgesia (PCA) using
Von Frey hair Test | measure at post-operative day 1, 9AM, before intervention; and post-operative day 2, 5PM, after intervention
  1. Pain, as assessed by von Frey hair Test at each wound sites
  2. Measure at post-operative day 1, 9AM, before intervention; and post-operative day 2, 5PM, after intervention
Vital signs | measure during whole admission, an average of 7 days
  1. Measure at every 9AM, 1PM, 5PM and 9PM
  2. Including blood pressure, heart rate, breath rate, body temperature
Questionnaire | measure before discharge, an average at post operative day 5
  1. Including quality control of acupuncture, discomfort and satisfaction during whole admission, an average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yu Lu, MD, Principal Investigator — Division of thoracic surgery, China medical university hospital, Taiwan
Locations (1):
- Division of thoracic surgery, China medical university hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leaver HA, Craig SR, Yap PL, Walker WS. Lymphocyte responses following open and minimally invasive thoracic surgery. Eur J Clin Invest. 2000 Mar;30(3):230-8. doi: 10.1046/j.1365-2362.2000.00622.x. PMID 10692000
- [Background] Rizk NP, Ghanie A, Hsu M, Bains MS, Downey RJ, Sarkaria IS, Finley DJ, Adusumilli PS, Huang J, Sima CS, Burkhalter JE, Park BJ, Rusch VW. A prospective trial comparing pain and quality of life measures after anatomic lung resection using thoracoscopy or thoracotomy. Ann Thorac Surg. 2014 Oct;98(4):1160-6. doi: 10.1016/j.athoracsur.2014.05.028. Epub 2014 Jul 31. PMID 25086945
- [Background] Mulder DS. Pain management principles and anesthesia techniques for thoracoscopy. Ann Thorac Surg. 1993 Sep;56(3):630-2. doi: 10.1016/0003-4975(93)90933-9. PMID 8379756
- [Background] Kim JA, Kim TH, Yang M, Gwak MS, Kim GS, Kim MJ, Cho HS, Sim WS. Is intravenous patient controlled analgesia enough for pain control in patients who underwent thoracoscopy? J Korean Med Sci. 2009 Oct;24(5):930-5. doi: 10.3346/jkms.2009.24.5.930. Epub 2009 Sep 23. PMID 19794994
- [Background] Lin JG, Chen WL. Acupuncture analgesia: a review of its mechanisms of actions. Am J Chin Med. 2008;36(4):635-45. doi: 10.1142/S0192415X08006107. PMID 18711761
- [Background] Lu KW, Hsu CK, Hsieh CL, Yang J, Lin YW. Probing the Effects and Mechanisms of Electroacupuncture at Ipsilateral or Contralateral ST36-ST37 Acupoints on CFA-induced Inflammatory Pain. Sci Rep. 2016 Feb 24;6:22123. doi: 10.1038/srep22123. PMID 26906464
- [Background] Wang B, Tang J, White PF, Naruse R, Sloninsky A, Kariger R, Gold J, Wender RH. Effect of the intensity of transcutaneous acupoint electrical stimulation on the postoperative analgesic requirement. Anesth Analg. 1997 Aug;85(2):406-13. doi: 10.1097/00000539-199708000-00029. PMID 9249122
- [Background] Kotani N, Hashimoto H, Sato Y, Sessler DI, Yoshioka H, Kitayama M, Yasuda T, Matsuki A. Preoperative intradermal acupuncture reduces postoperative pain, nausea and vomiting, analgesic requirement, and sympathoadrenal responses. Anesthesiology. 2001 Aug;95(2):349-56. doi: 10.1097/00000542-200108000-00015. PMID 11506105
- [Background] Langenbach MR, Aydemir-Dogruyol K, Issel R, Sauerland S. Randomized sham-controlled trial of acupuncture for postoperative pain control after stapled haemorrhoidopexy. Colorectal Dis. 2012 Aug;14(8):e486-91. doi: 10.1111/j.1463-1318.2012.02984.x. PMID 22330010
- [Background] Sim CK, Xu PC, Pua HL, Zhang G, Lee TL. Effects of electroacupuncture on intraoperative and postoperative analgesic requirement. Acupunct Med. 2002 Aug;20(2-3):56-65. doi: 10.1136/aim.20.2-3.56. PMID 12216602
- [Background] Lin JG, Lo MW, Wen YR, Hsieh CL, Tsai SK, Sun WZ. The effect of high and low frequency electroacupuncture in pain after lower abdominal surgery. Pain. 2002 Oct;99(3):509-514. doi: 10.1016/S0304-3959(02)00261-0. PMID 12406527
- [Background] Wang RR, Tronnier V. Effect of acupuncture on pain management in patients before and after lumbar disc protrusion surgery--a randomized control study. Am J Chin Med. 2000;28(1):25-33. doi: 10.1142/S0192415X00000052. PMID 10794114
- [Background] Ward U, Nilsson UG. Acupuncture for postoperative pain in day surgery patients undergoing arthroscopic shoulder surgery. Clin Nurs Res. 2013 Feb;22(1):130-6. doi: 10.1177/1054773812454136. Epub 2012 Jul 27. PMID 22843248
- [Background] Coura LE, Manoel CH, Poffo R, Bedin A, Westphal GA. Randomised, controlled study of preoperative electroacupuncture for postoperative pain control after cardiac surgery. Acupunct Med. 2011 Mar;29(1):16-20. doi: 10.1136/aim.2010.003251. PMID 21383391
- [Background] Gilbey P, Bretler S, Avraham Y, Sharabi-Nov A, Ibrgimov S, Luder A. Acupuncture for posttonsillectomy pain in children: a randomized, controlled study. Paediatr Anaesth. 2015 Jun;25(6):603-9. doi: 10.1111/pan.12621. Epub 2015 Feb 7. PMID 25661270
- [Background] Deng G, Rusch V, Vickers A, Malhotra V, Ginex P, Downey R, Bains M, Park B, Rizk N, Flores R, Yeung S, Cassiletha B. Randomized controlled trial of a special acupuncture technique for pain after thoracotomy. J Thorac Cardiovasc Surg. 2008 Dec;136(6):1464-9. doi: 10.1016/j.jtcvs.2008.07.053. PMID 19114190